CLINICAL TRIAL: NCT04355767
Title: Clinical-trial of COVID-19 Convalescent Plasma in Outpatients
Brief Title: Convalescent Plasma in Outpatients With COVID-19
Acronym: C3PO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Strategies to Innovate EmeRgENcy Care Clinical Trials Network (Network); University of Pittsburgh (Other); Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C3PO; 1OT2HL156812-01 (NIH)
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Results first posted 2021-10-19 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (Experimental): Participants receive 1 unit of convalescent plasma.
  Interventions: Biological: Convalescent Plasma
- Placebo (Placebo Comparator): Participants receive 1 unit of saline with multivitamin.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: Convalescent Plasma — SARS-CoV-2 convalescent plasma with neutralizing SARS-CoV2 antibodies titers of ≥1:160 administered via intravenous (IV) infusion.
  Arms: Convalescent Plasma
Biological: Saline — Saline with multivitamin administered via intravenous (IV) infusion..
  Arms: Placebo

SUMMARY:
The overarching goal of this project is to confirm or refute the role of passive immunization as a safe and efficacious therapy in preventing the progression from mild to severe/critical COVID-19 illness and to understand the immunologic kinetics of anti-SARS-CoV-2 antibodies after passive immunization.The primary objective is to determine the efficacy and safety of a single dose of convalescent plasma (CP) for preventing the progression from mild to severe COVID-19 illness. The secondary objective is to characterize the immunologic response to CP administration.

This study will enroll adults presenting to the emergency department (ED) with mild, symptomatic, laboratory-confirmed COVID-19 illness, who are at high risk for progression to severe/critical illness, but who are clinically stable for outpatient management at randomization.

ELIGIBILITY:
Inclusion Criteria:

* One or more symptoms of COVID-19 illness and laboratory-confirmed SARS-CoV-2 infection
* Has at least one study defined risk factor for severe COVID-19 illness
* Clinical team deems stable for outpatient management without supplemental oxygen
* CP available at the site at the time of enrollment
* Duration of symptoms ≤ 7 days at ED presentation
* Informed consent from subject

Exclusion Criteria:

* Age less than 18 years
* Prisoner or ward of the state
* Presumed unable to complete follow-up assessments
* Prior adverse reaction(s) from blood product transfusion
* Receipt of any blood product within the past 120 days
* Treating clinical team unwilling to administer 300 ml fluid
* Enrollment in another interventional trial for COVID-19 illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2020-08-11 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifton W Callaway, MD, PhD, Principal Investigator — University of Pittsburgh; Valerie Durkalski-Mauldin, PhD, Principal Investigator — Medical University of South Carolina; Frederick Korley, MD, PhD, Principal Investigator — University of Michigan; Sharon Yeatts, PhD, Principal Investigator — Medical University of South Carolina; Robert Silbergleit, MD, Principal Investigator — University of Michigan; William Barsan, MD, Principal Investigator — University of Michigan; Kevin Schulman, MD, Study Director — Stanford University
Locations (53):
- United States (53):
  - Chandler Regional Medical Center, Chandler, Arizona
  - Valleywise Health Medical Center, Phoenix, Arizona
  - UCSD Health La Jolla, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Stanford University, Stanford, California
  - Harbor-UCLA Medical Center, Torrance, California
  - University of Colorado Hospital, Aurora, Colorado
  - UF Health Shands Hospital, Gainesville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Illinois Hospital, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - University of Louisville Hospital, Louisville, Kentucky
  - Maine Medical Center, Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Sinai-Grace Hospital, Detroit, Michigan
  - Spectrum Health Hospitals Butterworth Hospital, Grand Rapids, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - William Beaumont Hospital-Troy, Troy, Michigan
  - HealthPartners Methodist Hospital, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Barnes Jewish Hospital, St Louis, Missouri
  - Cooper University Hospital, Camden, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - SUNY Downstate Medical Center, Brooklyn, New York
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - William P. Clements Jr. University Hospital, Dallas, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - Froedtert Hospital, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The complete de-identified patient data set will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available indefinitely.
Access Criteria: Data requests will be managed by National Heart, Lung, and Blood Institute (NHLBI).
URL: https://biodatacatalyst.nhlbi.nih.gov/

REFERENCES:
- [Result] Korley FK, Durkalski-Mauldin V, Yeatts SD, Schulman K, Davenport RD, Dumont LJ, El Kassar N, Foster LD, Hah JM, Jaiswal S, Kaplan A, Lowell E, McDyer JF, Quinn J, Triulzi DJ, Van Huysen C, Stevenson VLW, Yadav K, Jones CW, Kea B, Burnett A, Reynolds JC, Greineder CF, Haas NL, Beiser DG, Silbergleit R, Barsan W, Callaway CW; SIREN-C3PO Investigators. Early Convalescent Plasma for High-Risk Outpatients with Covid-19. N Engl J Med. 2021 Nov 18;385(21):1951-1960. doi: 10.1056/NEJMoa2103784. Epub 2021 Aug 18. PMID 34407339
- See also: SIREN Network — https://siren.network/
- See also: Statistical Design and Analysis Plan for Sequential Parallel-Group RCT for COVID-19 (Harrell and Lindsell, 2020) — http://hbiostat.org/proj/covid19/bayesplan.html
- Available data/document: Individual Participant Data Set — https://biodatacatalyst.nhlbi.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 48 hospital emergency departments in 21 states.
Groups:
- Convalescent Plasma: Participants receive 1 unit of convalescent plasma (with neutralizing SARS-CoV2 antibodies) administered via intravenous (IV) infusion.
- Placebo: Participants receive 1 unit of saline with multivitamin administered via intravenous (IV) infusion.
Period: Overall Study
Arm/Group | Convalescent Plasma | Placebo
Started | 257 | 254
Intention-to-treat Population | 257 | 254
Had Data for 15-day Outcome | 257 | 254
Completed | 250 | 251
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Death | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Convalescent Plasma | Placebo | Total
Number analyzed (Participants) | 257 | 254 | 511
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 54 [42 to 62] | 54 [40 to 62] | 54 [41 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 139 | 274
  Male | 122 | 115 | 237
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 83 | 73 | 156
  Not Hispanic or Latino | 170 | 179 | 349
  Unknown or Not Reported | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 8 | 10 | 18
  Black | 49 | 54 | 103
  Other | 28 | 25 | 53
  White | 172 | 165 | 337
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 257 | 254 | 511
Eligibility risk factor [Count of Participants; unit: Participants]
  Age .50 yr | 155 | 155 | 310
  Body-mass index ≥30 | 152 | 150 | 302
  Hypertension | 105 | 111 | 216
  Current or former tobacco use | 81 | 71 | 152
  Diabetes mellitus | 76 | 66 | 142
  COPD or asthma | 56 | 68 | 124
  Coronary artery disease | 28 | 23 | 51
  Immunosuppression | 33 | 17 | 50
  Chronic lung disease | 16 | 15 | 31
  Chronic kidney disease | 16 | 12 | 28
  Congestive heart disease | 9 | 11 | 20
  Currently pregnant | 3 | 3 | 6
  Organ transplant recipient | 5 | 0 | 5
  Active cancer | 2 | 2 | 4
  Sickle-cell disease | 1 | 0 | 1
Number of eligibility risk factors [Count of Participants; unit: Participants]
  1 | 51 | 66 | 117
  3 | 65 | 65 | 130
  ≥3 | 141 | 123 | 264
Other coexisting illness [Count of Participants; unit: Participants]
  Current or former alcohol abuse | 20 | 16 | 36
  Current or former drug abuse | 18 | 17 | 35
  Thromboembolic disorder | 15 | 10 | 25
  Liver disease | 12 | 6 | 18
  Other hematologic disorder | 9 | 8 | 17
Symptom duration before randomization [Median (Inter-Quartile Range); unit: days] | 4 [2 to 5] | 3 [2 to 5] | 4 [2 to 5]
Interval between randomization and infusion [Median (Inter-Quartile Range); unit: minutes] | 92 [76 to 128] | 69 [48 to 96] | 81 [63 to 110]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Disease Progression (Intention-to-treat Population)
Description: Disease progression defined as death or hospital admission or seeking emergency or urgent care within 15 days of randomization.
Time Frame: 15 days
Population: Intention-to-treat population included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Placebo
Number analyzed (Participants) | 257 | 254
Participants
  Patients with a disease-progression event | 77 | 81
  Hospital admission for any reason | 51 | 56
  Seeking emergency or urgent care | 25 | 25
  Death without hospitalization | 1 | 0
Statistical Analysis 1: Comparison: Convalescent Plasma vs Placebo; Analysis is of patients with a disease-progression event. The trial required a sample size of 900 patients to detect an absolute between-group difference of 10 percentage points (the minimum difference that we considered to be clinically important) with a power of 85%; Test type: Superiority; A Bayesian framework was used to calculate a risk difference of 1.9 percentage points (placebo group minus convalescent-plasma group) with a 95% credible interval of -6.0 to 9.8. The posterior probability of superiority was calculated to be 0.68. Efficacy was defined as a posterior probability of 0.975 or more that the proportion of patients with outcome events was higher in the placebo group
Statistical Analysis 2: Comparison: Convalescent Plasma vs Placebo; Analysis is of patients with a disease-progression event; Test type: Superiority; Risk Difference (RD) = 2.2, 95% CI 2-sided [-5.9 to 10.4] — Risk difference after adjustment for age, sex, symptom duration

2. Primary Outcome: Number of Patients With Disease Progression (Per-protocol Population)
Description: as for outcome 1
Time Frame: 15 days
Population: Per-protocol population included all the patients who had undergone randomization after the exclusion of those who did not receive the assigned trial product, had an identified eligibility violation, or had a disease-progression event before the initiation of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Placebo
Number analyzed (Participants) | 246 | 251
Participants
  Patients with a disease-progression event | 71 | 80
  Hospital admission for any reason | 47 | 55
  Seeking emergency or urgent care | 24 | 25
  Death without hospitalization | 0 | 0
Statistical Analysis 1: Comparison: Convalescent Plasma vs Placebo; Analysis is of patients with a disease-progression event; Test type: Superiority; A Bayesian framework was used to calculate a risk difference of 3.0 percentage points (placebo group minus convalescent-plasma group) with a 95% credible interval of -4.9 to 10.8. The posterior probability of superiority was calculated to be 0.76. Efficacy was defined as a posterior probability of 0.975 or more that the proportion of patients with outcome events was higher in the placebo group

3. Secondary Outcome: Worst Severity Rating on the WHO COVID Ordinal Scale for Clinical Improvement During the 30 Days Following Randomization
Description: This scale was developed by a special World Health Organization (WHO) committee for quantifying COVID-19 illness severity.
  * 1 = Not hospitalized without limitation in activity (no symptoms)
  * 2 = Not hospitalized with limitation in activity (continued symptoms)
  * 3 = Hospitalized not on supplemental oxygen
  * 4 = Hospitalized on supplemental oxygen by mask or nasal prongs
  * 5 = Hospitalized on non-invasive ventilation or high flow nasal cannula
  * 6 = Hospitalized, intubated and mechanically ventilated
  * 7 = Hospitalized, intubated, mechanically ventilated and requiring additional organ support (pressors, renal replacement therapy)
  * 8 = Death
Time Frame: 30 days
Population: Participants with available data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Placebo
Number analyzed (Participants) | 250 | 248
Participants
  Severity rating 1 | 55 | 55
  Severity rating 2 | 141 | 133
  Severity rating 3 | 12 | 17
  Severity rating 4 | 28 | 35
  Severity rating 5 | 6 | 5
  Severity rating 6 | 1 | 0
  Severity rating 7 | 2 | 2
  Severity rating 8 | 5 | 1

4. Secondary Outcome: Number of Patients With Worsening of Symptoms at Day 15 as a Measure of Time to Disease Progression
Description: Assessed on the COVID Outpatient Ordinal Outcome Scale censored at 15 days after randomization. Scale provides more granular detail for outpatients than the WHO scale (adapted from Harrell and Lindsell, 2020). Worsening of symptoms is defined as any subject admitted to the hospital (level 1), seen in the emergency room (level 2), a patient who reports increased symptoms of 2 levels on the scale over a 24 hour period, or a patient who reports increased symptoms of 1 level observed for a 48 hour period.
  COVID Outpatient Ordinal Outcomes Scale
  * 1 = patient requires care in the hospital
  * 2 = patient requires care in the emergency department or urgent care
  * 3 = patient at home with symptoms rated as moderate (defined as fever, shortness of breath, abdominal pain)
  * 4 = patient at home with symptoms rated as mild (defined as afebrile, constitutional symptoms (flu-like illness) without shortness
  * 5 = patient in their usual state of health
Time Frame: 15 days
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Placebo
Number analyzed (Participants) | 257 | 254
Participants | 107 | 116
Statistical Analysis 1: Comparison: Convalescent Plasma vs Placebo; Test type: Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.69 to 1.17]

5. Secondary Outcome: Number of Hospital-free Days During the 30 Days Following Randomization
Time Frame: 30 days
Population: Intention-to-treat population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Convalescent Plasma | Placebo
Number analyzed (Participants) | 257 | 254
days | 28.3 (4.9) | 28.6 (3.6)
Statistical Analysis 1: Comparison: Convalescent Plasma vs Placebo; Test type: Other; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.4 to 1.1]

6. Secondary Outcome: All-cause Mortality
Time Frame: Assessed at 30 days
Population: Intention-to-treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Convalescent Plasma | Placebo
Number analyzed (Participants) | 257 | 254
Participants | 5 | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Convalescent Plasma | Placebo
All-Cause Mortality (participants affected / at risk) | 5/257 | 1/254
Serious Adverse Events (participants affected / at risk) | 59/257 | 64/254
Other Adverse Events (participants affected / at risk) | 51/257 | 35/254
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Plasma (N=257) | Placebo (N=254)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Influenza like illness (General disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 30 | 39
Septic shock (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 0
Oesophagoscopy (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
End stage renal disease, could not get outpatient dialysis (Renal and urinary disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Hypotension (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Convalescent Plasma (N=257) | Placebo (N=254)
Vertigo (Ear and labyrinth disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Chest pain (General disorders) | 3 | 7
Fatigue (General disorders) | 2 | 0
Infusion site extravasation (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 7 | 1
Sinusitis (Infections and infestations) | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 11 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Coronavirus test positive (Investigations) | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 1
Migraine (Nervous system disorders) | 3 | 1
Presyncope (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This study did not meet its maximum sample size of 900 participants due to a planned interim analysis that indicated that it was unlikely that there would be a difference in the rate of disease progression between the two groups if continued to the planned sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/67/NCT04355767/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT04355767/ICF_000.pdf